CLINICAL TRIAL: NCT05889104
Title: The Effect of Progressive Loading Protocol on Bone Mineral Density and Quality of Life in Osteoporotic Patients.
Brief Title: Effect of Progressive Loading Protocol on Bone Mineral Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Saeed Mufleh, Senior Physiotherapist, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PLP on Bone Mineral in OR Pt.
Record Dates: First submitted 2023-05-11; First posted 2023-06-05 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis
Keywords: Quality of life; Bone Mineral
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Progressive Loading Group (PLG) (Experimental): using Progressive Loading protocol.
  Interventions: Other: Progressive Loading Protocol (PLP):
- TheControl Group (CG) (Other): using a randomization program
  Interventions: Other: Randomization Program

INTERVENTIONS:
Other: Randomization Program — The subjects in the Control Group will undergo twelve weeks of low impact Aerobics Training along with a health awareness program
  Arms: TheControl Group (CG)
Other: Progressive Loading Protocol (PLP): — he subjects in the Progressive Loading Group will undergo 4-7 days of moderate to high impact loading activities per week.
  Arms: The Progressive Loading Group (PLG)

SUMMARY:
The aims of this study are to examine the effects of Progressive Loading Exercises Protocol on Bone Mineral Density in osteoporotic patient's well-being and quality of life before a fracture occurs in order to create remedies. In addition, the available data from health research and clinical studies on osteoporosis will be evaluated for their impact on patient well-being and quality of life, providing an up-to-date and comprehensive overview of evidence-based treatments.

DETAILED DESCRIPTION:
Progressive Loading Protocol (PLP): The subjects in the Progressive Loading Group will undergo 4-7 days of moderate to high impact loading activities per week for the duration of 6 weeks. The PLP is adapted and modified based on Exercise and Sports Science Australia (ESSA) position statement on exercise prescription for the prevention and management of Osteoporosis. The participants in the progressive loading group will perform vertical and multidirectional jumping, bounding, hopping, skipping rope, drop jumps and bench stepping. The weight bearing intensity will be progressed by increasing heights for activities such as bounding and drop jumping, adding weighted vests and changing directions. To prevent the risk of injury, the participants would be instructed to avoid the loaded spine flexion or twisting movements of the spine. Frail individuals should be supervised and exercised within reach of a railing or other stable support.

Intensity: Moderate-to-high weight bearing impact loads (>2 times body weight) that are progressive, novel, and multidirectional, within the limits of pain, increasing as tolerated.

Frequency: 4-7 days per week

Sets/Repetitions: Aim to work up to 50 repetitions over time (5 sets of 10 repetitions with 1-2 min rest between sets)

The subjects in the Control Group will undergo twelve weeks of low impact Aerobics Training along with a health awareness program..

ELIGIBILITY:
Inclusion Criteria:

* Subject with history of diabetes, hypertension

Exclusion Criteria:

* Subject with history of kidney diseases, cardiopulmonary diseases, thrombosis, hyperprolactinemia, spondylolisthesis, back/leg deformities or surgeries, osteoarthritis, pacemakers, implants of the lower extremity and spine, tumors, migraines, or having any other diseases that affect bone metabolism or neuromuscular performance.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Measuring the result of change by Dual energy x ray absorptiometry (DXA) During the Intervention | At the start of the intervention, then the measurement is done again after six weeks..
  to measure bone mineral density (BMD) at the spine and hip region. and hip regio

CONTACTS AND LOCATIONS:
Overall Officials: SAEED MUFLEH ALNASSER, MSc, Study Chair — Armed Forces Hospital
Locations (1):
- Armed Forces Hospital, Khamis Mushait, 'Asir Region, Saudi Arabia